CLINICAL TRIAL: NCT04155437
Title: Assessing the Feasibility of Integrating a Package of Maternal Nutrition Interventions Into Antenatal Care Services in Burkina Faso: A Cluster-Randomized Evaluation
Brief Title: Assessing the Feasibility of Integrating a Package of Maternal Nutrition Interventions Into Antenatal Care Services in Burkina Faso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: AFRICSanté (Other); FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHND-19-1052
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Maternal Dietary Diversity; Iron-Folic Acid Supplementation; Early Initiation of Breastfeeding
Keywords: maternal nutrition; antenatal care; Burkina Faso

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A&T intervention areas: intensified maternal nutrition behavior change interventions during antenatal care delivered through government health facilities.
  Interventions: Behavioral: Health Facility Level Interventions; Behavioral: Community Level Interventions; Behavioral: Health System Level Interventions
- Control (No Intervention): Comparison areas: standard antenatal care services delivered at government health facilities.

INTERVENTIONS:
Behavioral: Health Facility Level Interventions — * Intensified counseling on maternal dietary diversity and quality using job aids
  * Counseling on purpose of IFA supplementation, managing side effects, and importance of adherence to daily consumption
  * Distribution/prescription of IFA tablets at each ANC visit
  * Use of pill card/reminders for pregnant women and their spouses
  * Monthly IFA tablet stock monitoring to assure sufficient supplies
  * Measurement of weight gain during each ANC visit and advise on healthy weight gain
  * Checks for functioning scales and use of monitoring sheets
  * Intensified counseling on early initiation of breastfeeding and exclusive breastfeeding using job aids
  * Reminder on importance of early ANC attendance and 4+ visits
  Arms: Intervention
Behavioral: Community Level Interventions — * Advocacy among community leaders (traditional and religious leaders, local associations, etc.) about ANC
  * Gatherings among grandmothers, husbands, and other influencers about ANC and their roles
  * Promotion of ANC service utilisation and the importance of early ANC visit during the first trimester.
  * Early identification of pregnant women
  * Support women's group discussions
  * 2-3 home visits per pregnant woman by community health workers (Agent de santé a base communautaire; ASBC) which will include counseling on diet quality, breastfeeding, importance on adherence to daily IFA consumption and side effect management, etc.
  Arms: Intervention
Behavioral: Health System Level Interventions — * Training on nutrition interventions during ANC for all ANC providers and community health workers
  * Semi-annual supervision by the Regional Health Directorate (Direction Regionale de la Santé; DRS)
  * Quarterly supportive supervision of health facility staff by the health district management team
  * Monthly supportive supervision of ASBCs
  * Monthly review between health facilities and ASBCs
  * Training and use of data registers
  * Training and use of mother's cards to record up to 8 ANC visits and nutrition services
  * Training on data utilization to improve coverage and quality
  Arms: Intervention

SUMMARY:
Alive & Thrive (A&T) is an initiative that supports the scaling up of nutrition interventions to save lives, prevent illnesses, and contribute to healthy growth and development through improved maternal nutrition, breastfeeding and complementary feeding practices. In Burkina Faso, A&T developed an intensive package of maternal nutrition interventions to be integrated into existing ANC services delivered through government health facilities that align with the latest global evidence. These included intensified counseling and support on dietary diversity and quality during pregnancy, iron-folic acid (IFA) supplements consumption, importance of ANC and increasing the number of visits, adequate weight-gain monitoring, and early initiation of and exclusive breastfeeding. The evaluation used a two-arm cluster-randomized, non-masked trial design, consisting of two cross-sectional surveys of pregnant and recently delivered women (i.e. with a child under 6 months of age) in 2019 and 2021.

DETAILED DESCRIPTION:
Routine antenatal care (ANC) offers opportunities to receive a broad range of health promotion and prevention services including support for adequate nutritional care for pregnant women and their newborns, and any required medical treatment. In 2016, World Health Organization (WHO) updated its guidelines on ANC with a high priority placed on nutrition interventions. These guidelines also recommended increasing the number of ANC from at least four to eight contacts to improve women's positive experience of care and to reduce perinatal morbidity and mortality. Following these new recommendations, the government of Burkina Faso is working with WHO and other partners to revise the national guidelines on ANC and test elements of the essential core package of routine ANC needed by women throughout pregnancy.

A&T Burkina Faso, developed an intensive package of maternal nutrition interventions to be integrated into existing ANC services delivered through government health facilities that align with the latest global evidence. These included intensified counseling and support on dietary diversity and quality during pregnancy, iron-folic acid (IFA) supplements consumption, importance of ANC and increasing the number of visits, adequate weight-gain monitoring, and early initiation of and exclusive breastfeeding. IFPRI tested the feasibility of the behavior-change interventions and examined their impacts on pregnant women's health and nutrition practices and breastfeeding practices of recently delivered women, compared with standard antenatal care services provided in control areas.

The study was designed as a two-arm cluster-randomized, non-masked trial, consisting of two cross-sectional surveys at baseline and endline. The unit of randomization was the health and social promotion center (CSPS, Centre de Santé et de Promotion Social in French) catchment area. 40 CSPS in Boucle du Mouhoun and 40 CSPS in Hauts-Bassins were randomly assigned to intervention/control. A baseline cluster/facility-level and household survey took place in November-December 2019. Soon after the completion of the baseline survey, the interventions were implemented at the CSPS and villages within the intervention areas for approximately 10 months (less than 1 year, caused by brief service interruptions in March-April 2020 due to the COVID-19 pandemic). The endline survey took place in January-March 2021.

The overall study objective is to evaluate the feasibility of integrating locally relevant maternal nutrition interventions into ANC services provided by the government health system and their impact on diet quality and quantity and utilization of nutrition interventions during pregnancy.

The implementation research study addresses three research questions:

1. What are the program impacts on maternal nutrition practices: (1) consumption of diversified foods and adequate intake of micronutrient, protein and energy compared to recommended intakes; (2) consumption of IFA supplements during pregnancy; and (3) early breastfeeding practices?
2. Can the coverage and utilization of key nutrition interventions (maternal nutrition counseling, weight gain monitoring, distribution of and counseling on IFA supplementation, and breastfeeding counseling) and number of ANC contacts be improved through health system strengthening and nutrition-focused social and behavior change communication (SBCC; interpersonal communication and community mobilization) approaches?
3. What factors influenced integration and strengthening of maternal nutrition interventions into the government ANC service delivery platform?

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant or recently delivered with a child 0-5.9 months of age
* Residency in the health facility catchment area
* Informed consent

Exclusion Criteria:

* Age <15 years or >49 years

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 8110 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Dietary diversity during pregnancy | Approximately 16 months after baseline in a cross-sectional endline survey
  Mean number of food groups consumed by pregnant women on the day preceding the interview.
Minimum dietary diversity during pregnancy | Approximately 16 months after baseline in a cross-sectional endline survey
  Proportion of pregnant women who consumed 5 or more food groups on the day preceding the interview.
Consumption of iron-folic acid tablets during pregnancy | Approximately 16 months after baseline in a cross-sectional endline survey
  Mean number of IFA tablets consumed during last pregnancy by recently delivered women with a child 0-5.9 months of age.
Consumption of 90+ iron-folic acid tablets during pregnancy | Approximately 16 months after baseline in a cross-sectional endline survey
  Proportion of women who consumed 90+ IFA tablets during last pregnancy by recently delivered women with a child 0-5.9 months of age.

SECONDARY OUTCOMES:
Micronutrient, protein and energy adequacy during pregnancy | Approximately 16 months after baseline in a cross-sectional endline survey
  Proportion of pregnant women whose micronutrient, protein and energy intakes are equal to or above the dietary reference intake.
Early initiation of breastfeeding | Approximately 16 months after baseline in a cross-sectional endline survey
  Proportion of children aged 0-5.9 months who were breastfed within 1 hour of birth.
Use of ANC services during pregnancy | Approximately 16 months after baseline in a cross-sectional endline survey
  Total number of ANC visits and month of first ANC first during last pregnancy reported by recently delivered women with a child age 0-5.9 months.
Exposure to nutrition interventions during ANC | Approximately 16 months after baseline in a cross-sectional endline survey
  Proportion of recently delivered women with children 0-5.9 months of age who received nutrition interventions during their last pregnancy during ANC and in the community based on survey responses.
Women's knowledge of maternal nutrition and breastfeeding | Approximately 16 months after baseline in a cross-sectional endline survey
  Proportion of recently delivered women with children 0-5.9 months of age with correct knowledge of maternal nutrition and appropriate breastfeeding practices based on survey responses.
Health worker knowledge of IFA supplementation, dietary diversity, weight gain during pregnancy, and early and exclusive breastfeeding. | Approximately 16 months after baseline in a cross-sectional endline survey
  Proportion of Nurse-Midwives and community health workers (ASBCs) with correct knowledge of IFA supplementation, dietary diversity, weight gain during pregnancy and appropriate breastfeeding practices based on survey responses.
Availability of ANC service supports | Approximately 16 months after baseline in a cross-sectional endline survey
  Proportion of health facilities with ANC materials and equipment based on enumerator observation.

CONTACTS AND LOCATIONS:
Locations (1):
- International Food Policy Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
In compliance with donor open access policy requirements, fully anonymized datasets will be made publicly available one year after the end of the project. Metadata and other documentation of data collection procedures (such as the codebook, data collection instruments and interviewer guides/protocols) will also be made publicly available.
Supporting Information: Study Protocol, ICF
Time Frame: Fully anonymized datasets will be made publicly available one year after the end of the project.

REFERENCES:
- [Background] Hanson MA, Bardsley A, De-Regil LM, Moore SE, Oken E, Poston L, Ma RC, McAuliffe FM, Maleta K, Purandare CN, Yajnik CS, Rushwan H, Morris JL. The International Federation of Gynecology and Obstetrics (FIGO) recommendations on adolescent, preconception, and maternal nutrition: "Think Nutrition First". Int J Gynaecol Obstet. 2015 Oct;131 Suppl 4:S213-53. doi: 10.1016/S0020-7292(15)30034-5. No abstract available. PMID 26433230
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] WHO Recommendations on Antenatal Care for a Positive Pregnancy Experience. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK409108/ PMID 28079998
- [Background] Partnership for Maternal, Newborn and Child Health (PMNCH). 2006. Opportunities for Africa's newborns: Practical data, policy and programmatic support for newborn care in Africa. Edited by Joy Lawn and Kate Kerber. Cape Town: PMNCH.
- [Background] United Nations Children's Fund (UNICEF). 2016. The state of the world's children 2016: A fair chance for every child. New York: UNICEF.
- [Background] Alkema L, New JR, Pedersen J, You D; UN Inter-agency Group for Child Mortality Estimation; Technical Advisory Group. Child mortality estimation 2013: an overview of updates in estimation methods by the United Nations Inter-agency Group for Child Mortality Estimation. PLoS One. 2014 Jul 11;9(7):e101112. doi: 10.1371/journal.pone.0101112. eCollection 2014. PMID 25013954

DOCUMENTS (3):
  • Study Protocol (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT04155437/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04155437/SAP_001.pdf
  • Informed Consent Form (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT04155437/ICF_002.pdf